CLINICAL TRIAL: NCT03783819
Title: Effects of Hypericum Perforatum Oil on Promoting Skin Recovery in Different Human Skin Damage Models, Randomized Controlled Trial
Brief Title: Effects of Hypericum Perforatum Oil on Promoting Skin Recovery in Different Human Skin Damage Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2181-198-03-01-18-0058
Record Dates: First submitted 2018-12-17; First posted 2018-12-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Skin Recovery in Different Human Skin Damage Models
Keywords: Hypericum perforatum; Saint John's Wort; St. John's Wort
MeSH Terms: interventions — Hypericum extract LI 160; Ultraviolet Rays

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Active Comparator): One forearm will be treated with ointment containing Hypericum perforatum oil. Forearm (left or right) will be chosen according to randomization protocol.
  Interventions: Other: Hypericum perforatum oil; Procedure: SLS induced irritation; Procedure: Tape-stripping; Procedure: UV radiation; Procedure: Intact skin
- Placebo treatment (Placebo Comparator): Other forearm will be treated with placebo ointment. Forearm (left or right) will be chosen according to randomization protocol.
  Interventions: Other: Placebo; Procedure: SLS induced irritation; Procedure: Tape-stripping; Procedure: UV radiation; Procedure: Intact skin

INTERVENTIONS:
Other: Hypericum perforatum oil — Ointment containing Hypericum perforatum oil
  Arms: Active treatment
Other: Placebo — Ointment containing plant oils used in Hypericum perforatum oil production and dye
  Arms: Placebo treatment
Procedure: SLS induced irritation — 60 uL of 1% w/v sodium lauryl sulphate (SLS) will be applied to skin under occlusion by large Finn chamber for 24 hours as described in the guidelines by Standardization group of European Society of Contact Dermatitis. Procedure will be performed to specified skin sites, according to randomization protocol.
Procedure: Tape-stripping — Skin barrier disruption will be induced by tape-stripping. Procedure will be performed to specified skin sites, according to randomization protocol.
Procedure: UV radiation — UV radiation will be used to induce skin erythema and damage. Procedure will be performed to specified skin sites, according to randomization protocol.
Procedure: Intact skin — Healthy, intact skin. Procedure will be performed to specified skin sites, according to randomization protocol.

SUMMARY:
Saint John's wort (Hypericum perforatum) was recognised as a traditional, folk medicine used topically for the treatment of wounds, abrasions, burns, sunburns and inflammatory skin disorders.

Its use in wound healing could be justified with its anti-inflammatory, antimicrobial and astringent effects. It also stimulated tissue growth and cell differentiation, as one of Hypericum perforatum's main ingredients, hyperforin, was shown to activate TRPC6 channel which had been recognised as an activator of keratinocyte differentiation. Another potentially useful activities could be its inhibitory effects on epidermal Langerhans cells.

Furthermore, in vivo research showed its potential with improved wound healing in different rat models. Finally, several clinical studies were performed testing its effects in atopic dermatitis treatment, wound healing after caesarean section and episiotomy, as well as healing of post-surgical scalp wounds, bed sores and venous ulcers.

The aim of the study will be to determine the effectiveness of ointment containing Hypericum perforatum oil on promoting skin recovery in different human skin damage models on healthy volunteers, in comparison to placebo.

Chosen test sites will be the forearms. One forearm will be treated will the formulation containing Hypericum perforatum oil while the other will be treated with the placebo formulation. Four test sites will be marked on each forearm with skin barrier damage induced on three areas while the fourth will be left intact. Treated forearm and test sites sequence on forearms will be prospectively randomized (double randomization).

First skin damage model used in the trial will be sodium lauryl sulphate (SLS) induced irritation. The SLS solution will be placed on the skin of participants under the occlusion for 24 hours. Second model will be the tape-stripping procedure with defined TEWL value set as an endpoint. The final model will be damage by the UV radiation. UV irradiation will be performed under strict conditions with use of the necessary safety equipment. Only the defined test areas will be irradiated with the defined dose of radiation.

ELIGIBILITY:
Inclusion Criteria:

- young, healthy volunteers who gave written informed consent

Exclusion Criteria:

* skin disease, skin damage on measurement sites
* use of corticosteroids, antihistamines and immunomodulators a month prior the inclusion and during the trial
* use of drugs that may cause photosensitivity
* use of emollients three days prior the inclusion in the trial
* non-adherence to the trial protocol
* exposure to artificial and excessive natural UV radiation
* pregnancy and lactation
* skin cancer
* history of vitiligo, melasma and other pigmentation and photosensitivity disorders
* immunosuppression
* allergic or irritant reactions to the constituents of the two ointments (active and placebo) and similar chemicals (e.g. salicylic and benzoic acid)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss change | Assessments will be performed on 1st, 2nd, 3rd, 4th, 5th, 8th and 11th day of the trial (baseline measurements and change from baseline assessment).
  Tewameter will be used to assess skin barrier function as a measurement of the water loss (g/hm2).
Stratum corneum hydration change | Assessments will be performed on 1st, 2nd, 3rd, 4th, 5th, 8th and 11th day of the trial (baseline measurements and change from baseline assessment).
  Corneometer will be used to estimate skin dryness. It is a relative measurement and uses arbitrary units (AU).
Erythema change | Assessments will be performed on 1st, 2nd, 3rd, 4th, 5th, 8th and 11th day of the trial (baseline measurements and change from baseline assessment).
  Mexameter will be used to assess erythema. It is a relative measurement and uses arbitrary units (AU).
Melanin content change | Assessments will be performed on 1st, 2nd, 3rd, 4th, 5th, 8th and 11th day of the trial (baseline measurements and change from baseline assessment).
  Mexameter will be used to assess skin melanin content. It is a relative measurement and uses arbitrary units (AU).

CONTACTS AND LOCATIONS:
Overall Officials: Dario Leskur, MPharm, Principal Investigator — University of Split, School of Medicine
Locations (1):
- School of Medicine, Split, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wolfle U, Seelinger G, Schempp CM. Topical application of St. John's wort (Hypericum perforatum). Planta Med. 2014 Feb;80(2-3):109-20. doi: 10.1055/s-0033-1351019. Epub 2013 Nov 8. PMID 24214835
- [Background] Jaric S, Kostic O, Mataruga Z, Pavlovic D, Pavlovic M, Mitrovic M, Pavlovic P. Traditional wound-healing plants used in the Balkan region (Southeast Europe). J Ethnopharmacol. 2018 Jan 30;211:311-328. doi: 10.1016/j.jep.2017.09.018. Epub 2017 Sep 21. PMID 28942136
- [Background] Schempp CM, Winghofer B, Ludtke R, Simon-Haarhaus B, Schopf E, Simon JC. Topical application of St John's wort (Hypericum perforatum L.) and of its metabolite hyperforin inhibits the allostimulatory capacity of epidermal cells. Br J Dermatol. 2000 May;142(5):979-84. doi: 10.1046/j.1365-2133.2000.03482.x. PMID 10809859
- [Background] Davis J, Burr AR, Davis GF, Birnbaumer L, Molkentin JD. A TRPC6-dependent pathway for myofibroblast transdifferentiation and wound healing in vivo. Dev Cell. 2012 Oct 16;23(4):705-15. doi: 10.1016/j.devcel.2012.08.017. Epub 2012 Sep 27. PMID 23022034
- [Background] Suntar IP, Akkol EK, Yilmazer D, Baykal T, Kirmizibekmez H, Alper M, Yesilada E. Investigations on the in vivo wound healing potential of Hypericum perforatum L. J Ethnopharmacol. 2010 Feb 3;127(2):468-77. doi: 10.1016/j.jep.2009.10.011. Epub 2009 Oct 13. PMID 19833187
- [Background] Thandar Y, Gray A, Botha J, Mosam A. Topical herbal medicines for atopic eczema: a systematic review of randomized controlled trials. Br J Dermatol. 2017 Feb;176(2):330-343. doi: 10.1111/bjd.14840. Epub 2016 Nov 30. PMID 27373699
- [Background] Schempp CM, Windeck T, Hezel S, Simon JC. Topical treatment of atopic dermatitis with St. John's wort cream--a randomized, placebo controlled, double blind half-side comparison. Phytomedicine. 2003;10 Suppl 4:31-7. doi: 10.1078/1433-187x-00306. PMID 12807340
- [Background] Lavagna SM, Secci D, Chimenti P, Bonsignore L, Ottaviani A, Bizzarri B. Efficacy of Hypericum and Calendula oils in the epithelial reconstruction of surgical wounds in childbirth with caesarean section. Farmaco. 2001 May-Jul;56(5-7):451-3. doi: 10.1016/s0014-827x(01)01060-6. PMID 11482776
- [Background] Samadi S, Khadivzadeh T, Emami A, Moosavi NS, Tafaghodi M, Behnam HR. The effect of Hypericum perforatum on the wound healing and scar of cesarean. J Altern Complement Med. 2010 Jan;16(1):113-7. doi: 10.1089/acm.2009.0317. PMID 20064022
- [Background] Hajhashemi M, Ghanbari Z, Movahedi M, Rafieian M, Keivani A, Haghollahi F. The effect of Achillea millefolium and Hypericum perforatum ointments on episiotomy wound healing in primiparous women. J Matern Fetal Neonatal Med. 2018 Jan;31(1):63-69. doi: 10.1080/14767058.2016.1275549. Epub 2017 Feb 23. PMID 28027682
- [Background] Lauchli S, Hafner J, Wehrmann C, French LE, Hunziker T. Post-surgical scalp wounds with exposed bone treated with a plant-derived wound therapeutic. J Wound Care. 2012 May;21(5):228, 230, 232-3. doi: 10.12968/jowc.2012.21.5.228. PMID 22584740
- [Background] Tupker RA, Willis C, Berardesca E, Lee CH, Fartasch M, Agner T, Serup J. Guidelines on sodium lauryl sulfate (SLS) exposure tests. A report from the Standardization Group of the European Society of Contact Dermatitis. Contact Dermatitis. 1997 Aug;37(2):53-69. doi: 10.1111/j.1600-0536.1997.tb00041.x. PMID 9285167
- [Derived] Leskur D, Perisic I, Romac K, Susak H, Seselja Perisin A, Bukic J, Rusic D, Kladar N, Bozin B, Modun D. Comparison of mechanical, chemical and physical human models of in vivo skin damage: Randomized controlled trial. Skin Res Technol. 2021 Mar;27(2):208-216. doi: 10.1111/srt.12932. Epub 2020 Jul 20. PMID 32686217